CLINICAL TRIAL: NCT06650189
Title: Investigation of the Effect of Music on the Stress of Preterm Neonates Through Innovative Applications
Brief Title: Investigation of the Effect of muSic on the Stress of Preterm neONates Through innovATive Applications (SONATA)
Acronym: SONATA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Collaborators: General and Maternity Hospital of Athens Elena Venizelou (Other); Attikon Hospital (Other)
Responsible Party: Principal Investigator, Dimitra Metallinou, Assistant Professor, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 44834
Record Dates: First submitted 2024-09-27; First posted 2024-10-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-07

CONDITIONS: Premature Neonates
Keywords: preterm neonates; premature neonates; stress; salivary biomarkers; NICU; preterm infants; premature infants; music
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Preterm neonates will receive standard of care.
- Music intervention (Experimental): Preterm neonates will be exposed to recorded music intervention. Recorded music will be played through a portable Bluetooth speaker (3.1 watt) placed in the incubator, which will be activated and controlled via a smartphone.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — Recorded music created by a certified music therapist
  Arms: Music intervention

SUMMARY:
The goal of this prospective randomized clinical trial is to investigate the effect of music intervention on the stress of live born preterm neonates requiring admission to a Neonatal Intensive Care Unit, through the measurements of salivary biomarkers (hormones and proteins).

The main question it aims to answer is:

Can the daily music intervention reduce the stress levels created by the Neonatal Intensive Care Unit environment in preterm neonates?

Researchers will compare preterm neonates who will not be exposed to music intervention to investigate potential discrepancies in salivary stress biomarkers.

Participants will be exposed to recorded music for 5 consecutive days.

DETAILED DESCRIPTION:
Study Design In this prospective randomized controlled clinical trial, live born preterm neonates should have a stable clinical status at the time of study enrollment and therefore it is likely that some neonates will be enrolled after 5-7 days of admission. The allocation of neonates will be randomized in order to equalize the prognostic factors (confounding factors) between the groups. By using sequentially numbered envelopes, participants will be assigned to either intervention or control group by simple random allocation. In this way, researchers will avoid resulting in an unequal number of participants between the two groups. Researchers after obtaining parental informed consent, will request a sealed envelope from a staff member not involved in the study. The envelope will be opened and the allocation will be documented on a list, and signed by a member of the research team and a staff member as witness.

Participants The study will recruit preterm neonates. It has been estimated that with a sample of 35 neonates per group, the study will have more than 85% power to find differences in biomarkers between the intervention and control group, with an effect size equal to or greater than 0.72 and a significance level of 0.05.

Music Intervention Neonates will be placed in a closed incubator whose acoustic properties have been previously studied. Under the close surveillance of a team member, monitor alarms will be also silenced so as to decrease exposure to sudden and unpleasant auditory stimuli during music intervention. A mini portable speaker will be settled inside the incubator in appropriate conditions (volume level, distance e.t.c) for safety reasons.

Neonates allocated to the intervention group will be exposed to a specific piece of music, 30 minutes after feeding (if oral feeding exists), for a duration no more than 30 minutes that will be indicated from the certified music - therapist, experienced in working with preterm infants.

A questionnaire created by the research team will be administered to parents in order to investigate the neonate's prenatal exposure of music (as a fetus).

Data collection Biomarkers Salivary samples will be obtained from preterm neonates via salivette swabs. The polyester filter of the device will be partitioned into equal sections under sterile conditions to account for the small oral size of the neonates. One sample will be obtained before the music intervention and one sample 60 minutes after the music intervention, considering diurnal flow patterns. Saliva sampling is unlikely to cause stress or pain to the neonate. In the control group only one sample per day will be obtained within the same time period with the intervention group. Sample collection will be repeated in the same way everyday for 5 consecutive days. Each sample will be obtained before any stressful intervention (e.g. blood sampling, weighing, bathing, etc.). Furthermore, it is important to note that no other procedure that may reduce stress will take place simultaneously with music intervention (i.e. kangaroo care, gentle touching e.t.c) in order to interpret the effect of music more precisely. Saliva samples will be centrifuged very soon after collection and stored at -80oC until the laboratory analyses are performed. Measurements will be performed with cobas e411 automated analyzer or through ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Born between 28 - 36+6 weeks of gestation
* Absence of active infection including blood, urine, cerebrospinal fluid
* Absence of congenital and genetic disorders and chromosomal abnormalities
* Absence of nuclear jaundice
* Absence of endocrine disorders
* Absence of maternal use of illicit drugs prenatally
* Non - sedated neonates
* Positive bilateral transient evoked otoacoustic emissions
* Stable clinical condition
* Absence of brain injury

Exclusion Criteria:

* Diagnosis of brain injury after the enrollment
* Negative auditory brainstem response before discharge
* Clinical deterioration

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Salivary stress biomarker 1 - Hormone | From enrollment to 5 consecutive days.
  Concentration of the hormone (Units: μg/dL).
Salivary stress biomarker 2 - Enzyme | From enrollment to 5 consecutive days.
  Concentration of the enzyme (Units: U/L).
Salivary stress biomarker 3 - Protein | From enrollment to 5 consecutive days.
  Concentration of the protein (Units: μg/mL).

SECONDARY OUTCOMES:
Heart rate | Measured before, during, and after each music session daily. From enrollment to the end of intervention at 5 days.
  Measurement of heart rate (beats per minute).
Respiratory rate | Measured before, during, and after each music session daily. From enrollment to the end of intervention at 5 days.
  Measurement of respiratory rate (breaths per minute).
Oxygen saturation | Measured before, during, and after each music session daily. From enrollment to the end of intervention at 5 days.
  Measurement of oxygen saturation (percent).
Blood pressure | Measured before, during, and after each music session daily. From enrollment to the end of intervention at 5 days.
  Measurement of blood pressure (millimeters of mercury).
Weight | Measured daily, with cumulative weight gain assessed at the end of the 5 days.
  Measurement of weight (grams).
Head circumference | Day 1 and 5.
  Measurement of head circumference (centimeters).
Daily volume of milk consumed. | Feeding efficiency will be analyzed over the 5-day period.
  The volume of milk consumed will be recorded daily (milliliters).
Length of hospitalization | From the date of hospital admission to the date of discharge, assessed up to 6 months.
  Measurement of the length of hospitalization (days) in the neonatal intensive care unit.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - General and Maternity Hospital of Athens Elena Venizelou, Athens
  - Attikon General University Hospital, Chaïdári

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified individual participant data (IPD) may be shared upon reasonable request. Interested researchers may contact the Primary Investigator directly to request access. No external link or public repository will be provided.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Access to de-identified individual participant data (IPD) will be granted to qualified researchers upon reasonable request. Interested parties/research groups must submit a written proposal outlining the intended purpose, type of analysis to be conducted, and justification for access to the data.
  Data sharing will require the execution of a formal Data Sharing Agreement (DSA) to ensure data use is consistent with ethical and legal standards, including participant confidentiality and proper data handling.
  Requests will be reviewed by the Principal Investigator and/or a designated review panel. Evaluation will consider the scientific merit of the proposal, qualifications of the requesting researcher(s), and ethical considerations. Communication and submission of the proposal and signed DSA can be done via email to the Primary Investigator.
  Please contact the Primary Investigator directly for more information or to initiate a request.